CLINICAL TRIAL: NCT06394544
Title: Effects of Brazil Nut Supplementation on Inflammation, Oxidative Stress and Microbiota in Patients With Chronic Kidney Disease Undergoing Conservative Treatment
Brief Title: Effects of Brazil Nut Supplementation in Patients With Chronic Kidney Disease Undergoing Conservative Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DeniseMafraCPA
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Disease stage3; Chronic Kidney Disease Stage 3A; Chronic Kidney Disease Stage 3B; Chronic Kidney Disease stage4; Inflammation; Inflammatory Response; Oxidative Stress; Intestinal Microbiota
Keywords: Chronic Kidney Diseases; Conservative treatment; Inflammation; Oxidative stress; Intestinal microbiota; Brazil Nut
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — 2S albumin, brazil nut

STUDY DESIGN:
Intervention Model Description: A longitudinal, prospective clinical trial will be carried out with patients with CKD undergoing conservative treatment. Volunteers will be randomized into groups G1 and G2, and in the first stage, G1 will be in the intervention group and G2 in the control group. In the second stage, everyone will undergo washout and, in the third stage, a crossover between groups will be carried out, passing G2 to intervention and G1 to control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brazil nut (Experimental): Each patient will receive 30 units of Brazil nuts per month, to consume one nut/day for two months. The time and daily amount of nuts were based on the European Food Safety recommendation Authority (EFSA). The adequate value for selenium intake was determined by EFSA aiming at the maximum serum concentration of Selenoprotein P and glutathione peroxidase activity, reached between four and 10 weeks, with 70 µg/day; we consider that a Brazil nut can contain up to 400 µg of Se.
  The use of fresh nuts made it impossible to use a placebo with the same sensory characteristics. Then, in the control stage, volunteers will receive conventional conservative nutritional treatment, without nut supplementation.
  Interventions: Dietary Supplement: Brazil Nut
- Washout (No Intervention): Time T2 will be a washout period , so that residual effects between stages T1 and T3 are avoided.
- Crossover (No Intervention): the crossover between the groups will allow the same participant to be exposed, at different times, to the intervention stage and the control stage.

INTERVENTIONS:
Dietary Supplement: Brazil Nut — The intervention, for each participant, is estimated to last a total period of six months , which will be divided into three two-month stages, with data collection after each stage. Volunteers will be monitored to control possible side effects, doubts and check compliance. In addition, the telephone number and an email will be made available for contact during business hours, for possible clarifications.
  Arms: Brazil nut

SUMMARY:
The aim of this study is to evaluate the effects of Brazil nut supplementation on inflammation, oxidative stress and intestinal microbiota in patients with chronic kidney disease undergoing conservative treatment.

DETAILED DESCRIPTION:
Complications such as inflammation and oxidative stress are common in chronic kidney disease (CKD) and directly influence the rate of disease progression. Patients with CKD also have intestinal dysbiosis, which aggravates the inflammatory process and oxidative stress, forming a vicious circle between inflammation, oxidative stress and intestinal dysbiosis. Nutritional strategies try to alleviate this circle and Brazil nuts, rich in bioactive compounds, have already been proven effective in mitigating inflammation and oxidative stress in CKD patients on dialysis. However, to date, the effectiveness of Brazil nuts in patients with CKD in stages prior to dialysis (conservative treatment) has not been tested. The bioactive compounds in Brazil nuts are expected to contribute positively to the redox balance, reduction of inflammation and intestinal eubiosis in patients with CKD undergoing conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than three months of nutritional monitoring at the Renal Nutrition Outpatient Clinic of the Universidade Federal Fluminense (UFF), between stages G3a and G4, will be included, according to KDOQI 2020 guidelines, and authorized by the medical and nutritionist team.

Exclusion Criteria:

* Current use or in the last three months of antibiotics, anti-inflammatories and/or antioxidant supplements. Patients who are allergic, intolerant, or regularly ingest Brazil nuts; pregnant/lactating women, smokers; undergoing cancer treatment, HIV-positive, or with any clinical condition that compromises the accuracy of the intervention.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in antioxidants and anti-inflammatory biomarkers | 8 weeks
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers- nuclear receptor factor 2 (Nrf2), glutathioneperoxidase (GPx), heme oxygenase-1 (HO-1).

SECONDARY OUTCOMES:
Change in inflammatory biomarkers | 8 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers- factor nuclear kappa B (NFkB), interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-alpha).
Change in microbiota composition | 8 weeks
  DNA extraction from fecal samples will be carried out using the kit QIAamp DNA Stool Mini Kit.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Rodrigues, MS, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil